CLINICAL TRIAL: NCT05372367
Title: An Open-label Fixed Sequence Trial to Investigate the Potential Drug-drug Interaction When BI 907828 is Co-administered With an OATP1B1 and/or OATP1B3 Transporter Inhibitor or With a CYP3A4 Inhibitor in Patients With Various Solid Tumours
Brief Title: A Study in People With Advanced Cancer to Test Whether the Amount of BI 907828 in the Blood is Influenced by Taking an OATP Inhibitor or a CYP3 Inhibitor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1403-0004; 2021-006565-38 (EudraCT Number); 2024-514532-24-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2022-05-09; First posted 2022-05-12 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Solid Tumors
MeSH Terms: interventions — brigimadlin; Rifampin; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: OATP1B1/B3 inhibitor (Experimental)
  Interventions: Drug: BI 907828; Drug: Rifampicin
- Group 2: CYP3A4 inhibitor (Experimental)
  Interventions: Drug: BI 907828; Drug: Itraconazole

INTERVENTIONS:
Drug: BI 907828 — BI 907828
  Other Names: Brigimadlin
Drug: Rifampicin — Rifampicin
  Arms: Group 1: OATP1B1/B3 inhibitor
Drug: Itraconazole — Itraconazole
  Arms: Group 2: CYP3A4 inhibitor

SUMMARY:
This study is open for adults with advanced cancer (solid tumours). This is a study for people for whom previous treatment was not successful.

This study tests a medicine called BI 907828. BI 907828 is a so-called MDM2 inhibitor that is being developed to treat cancer. The purpose of this study is to find out whether the amount of BI 907828 in the blood is influenced by taking an OATP inhibitor or a CYP3 inhibitor. This study uses an OATP inhibitor called rifampicin and a CYP3 inhibitor called itraconazole. In clinical practice, rifampicin is used as an antibiotic. Itraconazole is used to treat fungal infections.

Participants are divided into 2 groups: a rifampicin group and an itraconazole group. Every participant takes BI 907828 as a tablet every 3 weeks. This is called a cycle.

* Rifampicin group: In addition to BI 907828, participants take 1 tablet of rifampicin in the second cycle.
* Itraconazole group: In addition to BI 907828, participants take itraconazole tablets for 20 days starting 1 week after the second cycle begins

Participants can stay in the study as long as they benefit from treatment and can tolerate it.

The doctors take blood samples from the participants to compare the amount of BI 907828 in the blood when it is taken alone and when participants also take rifampicin. Doctors also regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion criteria:

1. Age ≥18 and ≤70 years.
2. Signed and dated written informed consent in accordance with International Council on Harmonisation - Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial.
3. Male or female patients. Women of childbearing potential (WOCBP) and men able to father a child must be ready and able to use two medically acceptable methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly beginning at screening, during trial participation, and until 6 months and 12 days after last dose for women and 102 days after last dose for men. A list of contraception methods meeting these criteria is provided in the patient information.
4. Patients with histologically or cytologically confirmed diagnosis of advanced, non resectable and/or metastatic solid tumour.
5. Patient with either measurable or non-measurable disease. Non-evaluable disease is allowed.
6. Patient who has failed conventional treatment or for whom no therapy of proven efficacy exists or who is not eligible for established treatment options. Patient must have exhausted available treatment options known to prolong survival for their disease.
7. Patient has a tumour with either a known Tumor Protein p53 (TP53) wild type status, or unknown TP53 status, at the time of study entry.
8. Eastern Cooperative Oncology Group (ECOG) performance score 0 or 1. Further inclusion criteria apply.

Exclusion criteria:

1. Second malignancy currently requiring active therapy (except for hormonal /antihormonal treatment e.g. in prostate or breast cancer).
2. Chemo-, radio- immuno-, or molecular-targeted cancer-therapy within the past four weeks prior to start of BI 907828. This restriction does not apply to steroids, bisphosphonates hormonal / antihormonal treatment (e.g. in prostate or breast cancer).
3. Serious concomitant disease or medical condition which may affect compliance with trial requirements in the opinion of the Investigator.
4. Clinical evidence of active brain metastasis or leptomeningeal disease in the past 6 months prior to screening.
5. Active major infection requiring systemic treatment (antibacterial, antiviral, or antifungal therapy) at treatment start in this trial.
6. Known history of human immunodeficiency virus infection.
7. Patients with a history of Hepatitis C virus (HCV) infection who meet one or both of the following criteria:

   * Currently receiving curative antiviral treatment
   * HCV viral load is above the limit of quantification (HCV RNA positive)
8. Patients with chronic Hepatitis B virus (HBV) infection with active disease who meet the criteria for anti-HBV therapy (according to local / institutional standard) and who have not been treated with suppressive antiviral therapy prior to initiation of study treatment.

Further exclusion criteria apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-08-11 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2025-04-29 (Actual)

PRIMARY OUTCOMES:
Group 1: Area under the concentration-time curve of BI 907828 in plasma over the time interval from 0 to 24 hours (AUC 0-24) | up to 24 hours
Group 1: Maximum measured concentrations of BI 907828 in plasma (C max) | up to 15 days
Group 2: Area under the concentration-time curve of BI 907828 in plasma over the time interval from 0 to the last quantifiable data point (AUC 0-tz) | up to 15 days
Group 2: Maximum measured concentrations of BI 907828 in plasma (C max) | up to 15 days

SECONDARY OUTCOMES:
Group 1: Area under the concentration-time curve of BI 907828 in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | up to 15 days
Group 1: Area under the concentration-time curve of BI 907828 in plasma over the time interval from 0 to the last quantifiable data point (AUC 0-tz) | up to 15 days
Group 2: Area under the concentration-time curve of BI 907828 in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | up to 15 days

CONTACTS AND LOCATIONS:
Locations (7):
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Brussels
  - Wilrijk - HOSP GZA (St-Augustinus), Wilrijk
- Spain (5):
  - Hospital Quiron. I.C.U., Barcelona
  - Hospital Universitari Vall D Hebron, Barcelona
  - Fundación Jiménez Díaz, Madrid
  - CIO Clara Campal, Madrid
  - Hospital Quirónsalud Madrid, Madrid

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com